CLINICAL TRIAL: NCT02283268
Title: A Phase 3, Prospective, Multicenter Study to Evaluate Efficacy and Safety of Recombinant Von Willebrand Factor (rVWF) With or Without ADVATE in Elective Surgical Procedures in Subjects With Severe Von Willebrand Disease
Brief Title: Recombinant Von Willebrand Factor in Subjects With Severe Von Willebrand Disease Undergoing Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxalta now part of Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 071101; 2014-003575-38 (EudraCT Number)
Record Dates: First submitted 2014-10-27; First posted 2014-11-05 (Estimated); Results first posted 2017-08-31 (Actual); Last update posted 2021-05-19 (Actual); Status verified 2021-04

CONDITIONS: Von Willebrand Disease
MeSH Terms: conditions — von Willebrand Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Recombinant von Willebrand Factor (rVWF) (Experimental): Surgery participants treated with Recombinant von Willebrand Factor (rVWF)
  Interventions: Biological: Recombinant von Willebrand Factor (rVWF)

INTERVENTIONS:
Biological: Recombinant von Willebrand Factor (rVWF) — rVWF will be administered by intravenous bolus infusion. Participants planned for major surgery will undergo a baseline pharmacokinetic assessment prior to surgery. The peri- and postoperative substitution regimen will be individualized according to the PK results, intensity and duration of the hemostatic challenge, and the institution´s standard of care.

SUMMARY:
The purpose of the study is to assess the efficacy and safety of recombinant von Willebrand factor (rVWF) with or without ADVATE in major and minor elective surgical procedures in adult patients with hereditary severe von Willebrand disease (VWD).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of severe von Willebrand disease (VWD) as listed below and elective surgical procedure planned

  1. Type 1 (Von Willebrand factor : Ristocetin cofactor activity (VWF:RCo) <20 IU/dL), or
  2. Type 2A (as verified by multimer pattern), Type 2B (as diagnosed by genotype), Type 2N (FVIII:C<10% and historically documented genetics), Type 2M, or
  3. Type 3 (Von Willebrand factor antigen (VWF:Ag) ≤ 3 IU/dL)
* VWD with a history of requiring substitution therapy with von Willebrand factor (VWF) concentrate to control bleeding
* If type 3 VWD (VWF Antigen /VWF:Ag ≤ 3 IU/dL), participant has a medical history of at least 20 exposure days to VWF/FVIII coagulation factor concentrates (including cryoprecipitate or fresh frozen plasma)
* If type 1 or type 2 VWD, participant has a medical history of 5 exposure days or a past major surgery requiring VWF/FVIII coagulation factor concentrates (including cryoprecipitate or fresh frozen plasma)
* Participant is at least 18 years of age
* If female of childbearing potential, participant presents with a negative pregnancy test
* If applicable, participant agrees to employ adequate birth control measures for the duration of the study
* Participant is willing and able to comply with the requirements of the protocol

Exclusion Criteria:

* Diagnosis of pseudo VWD or another hereditary or acquired coagulation disorder (eg, qualitative and quantitative platelet disorders or elevated prothrombin time [PT] / international normalized ratio [INR] > 1.4)
* History or presence of a VWF inhibitor at screening
* History or presence of a factor VIII (FVIII) inhibitor with a titer ≥ 0.4 BU (Nijmegen-modified Bethesda assay ) or ≥ 0.6 BU (by Bethesda assay)
* Known hypersensitivity to any of the components of the study drugs, such as to mouse or hamster proteins
* Medical history of immunological disorders, excluding seasonal allergic rhinitis/conjunctivitis, mild asthma, food allergies or animal allergies
* Medical history of a thromboembolic event
* HIV positive with an absolute CD4 count < 200/mm3
* Platelet count < 100,000/mL
* Diagnosis of significant liver disease, as evidenced by, but not limited to, any of the following: serum alanine aminotransferase (ALT) 5 times the upper limit of normal; hypoalbuminemia; portal vein hypertension (eg. presence of otherwise unexplained splenomegaly, history of esophageal varices) or liver cirrhosis classified as Child B or C
* Diagnosis of renal disease, with a serum creatinine level ≥ 2 .5mg/dL
* Participant has been treated with an immunomodulatory drug, excluding topical treatment (eg, ointments, nasal sprays), within 30 days prior to signing the informed consent
* Participant is pregnant or lactating at the time informed content is obtained
* Participant has participated in another clinical study involving an investigational product (IP), other than rVWF with or without ADVATE, or investigational device within 30 days prior to enrollment or is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study. However, eligible patients participating in the rVWF Prophylaxis Study (071301) may be enrolled.
* Progressive fatal disease and/or life expectancy of less than 3 months
* Participant is identified by the investigator as being unable or unwilling to cooperate with study procedures
* Participant suffers from a mental condition rendering him/her unable to understand the nature, scope and possible consequences of the study and/or evidence of an uncooperative attitude
* Participant is in prison or compulsory detention by regulatory and/or juridical order
* Participant is a member of the study team conducting this study or in a dependent relationship with one of the study team members. Dependent relationships include close relatives (ie, children, partner/spouse, siblings, parents) as well as employees.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-04-01 (Actual); Primary Completion 2016-07-06 (Actual); Study Completion 2016-07-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (34):
- United States (12):
  - University of Colorado Hemophilia & Thrombosis Center, Aurora, Colorado
  - University of Miami, Jackson Memorial Hospital, Miami, Florida
  - Georgia Regents University, Augusta, Georgia
  - John Hopkins University, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Rutgers - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University Hospital, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Medical University of South Carolina (MUSC), Charleston, South Carolina
  - Blood Center of South East Wisconsin, Milwaukee, Wisconsin
- Australia (3):
  - Royal Adelaide Hospital, Adelaide, South Australia
  - The Perth Blood Institute, Nedlands, Western Australia
  - Fiona Stanley Hospital, Perth, Western Australia
- AKH - Medizinische Universität Wien, Vienna, Austria
- Fakultni nemocnice Ostrava, Ostrava, Czechia
- Universitätsmedizin der Johannes Gutenberg Universität Mainz, Mainz, Rhineland-Palatinate, Germany
- Italy (3):
  - Azienda Ospedaliero - Universitaria Careggi, Firenze (Florence)
  - Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan
  - Umberto I Policlinico di Roma, Universitá di Roma La Sapienza, Rome
- Erasmus Medisch Centrum, Rotterdam, Netherlands
- Russia (2):
  - Regional Budgetary State Healthcare Institution (SHI) "Regional Clinical Hospital", Barnaul
  - FSI Kirov Institute of Hematology and Blood Transfusion FMBA, Kirov
- Spain (2):
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitari i Politècnic La Fe, Valencia
- Taiwan (3):
  - Taichung Veterans General Hospital, Taichung
  - Tri-Service General Hospital, Taipei
  - National Taiwan University Hospital, Taipei
- Ege University Medical Faculty, Izmir, Turkey (Türkiye)
- SI Institute of Blood Pathology and Transfusion Medicine of NAMSU, Lviv, Ukraine
- United Kingdom (3):
  - Derriford Hospital, Plymouth, Devon
  - Royal Free Hospital, London, Greater London
  - Churchill Hospital, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment was conducted at 14 study sites in 10 countries (USA, Australia, Taiwan, Germany, Russia, Spain, Ukraine, United Kingdom, Italy, Turkey).
Pre-assignment Details: A total of 24 participants were enrolled (signed informed consent) and screened. Of these, 15 participants were treated with investigational product.
Period: Overall Study
Arm/Group | Recombinant Von Willebrand Factor (rVWF)
Started | 15
Completed | 14
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Recombinant Von Willebrand Factor (rVWF)
Number analyzed (Participants) | 15
Age, Continuous [Median (Full Range); unit: Years] | 40.0 [20.0 to 70.0]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Hemostatic Efficacy as Assessed by the Investigator (Hemophilia Physician)
Description: Hemostatic efficacy will be rated on a scale of excellent - good - moderate - none. Excellent: Intra-, and postoperative hemostasis achieved with rVWF with our without ADVATE was as good or better than that expected for the type of surgical procedure performed in a hemostatically normal subject. Good: Intra-, and postoperative hemostasis achieved with rVWF with or without ADVATE was probably as good as that expected for the type of surgical procedure performed in a hemostatically normal subject. Moderate: Intra-, and postoperative hemostasis with rVWF with or without ADVATE was clearly less than optimal for the type of procedure performed but was maintained without the need to change the rVWF concentrate. None: Participant experienced uncontrolled bleeding that was the result of inadequate therapeutic response despite proper dosing, necessitating a change of rVWF concentrate.
Time Frame: 24 hours after last peri-operative infusion or at completion of Day 14 (± 2 days) visit, whichever occurs earlier
Population: Number of participants with major, minor and oral surgery and number of participant with Von Willebrand Type 1, 2A, 2B, 2M and 3 do sum up to the overall number of participants analyzed. The full analysis data set, including all participants who received investigational product and have at least 1 hemostatic assessment, was used for analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Minor Surgery: All participants who underwent minor surgery.
- Major Surgery: All participants who underwent major surgery.
- Oral Surgery: All participants who underwent oral surgery.
- Von Willebrand Disease Type 1: All participants with von Willebrand Disease Type 1.
- Von Willebrand Disease Type 2A: All participants with von Willebrand Disease Type 2A.
- Von Willebrand Disease Type 2B: All participants with von Willebrand Disease Type 2B.
- Von Willebrand Disease Type 2M: All participants with von Willebrand Disease Type 2M.
- Von Willebrand Disease Type 3: All participants with von Willebrand Disease Type 3.
Arm/Group | Recombinant Von Willebrand Factor (rVWF) | Minor Surgery | Major Surgery | Oral Surgery | Von Willebrand Disease Type 1 | Von Willebrand Disease Type 2A | Von Willebrand Disease Type 2B | Von Willebrand Disease Type 2M | Von Willebrand Disease Type 3
Number analyzed (Participants) | 15 | 4 | 10 | 1 | 3 | 2 | 1 | 1 | 8
Participants
  Excellent | 11 | 4 | 7 | 0 | 2 | 1 | 1 | 0 | 7
  Good | 4 | 0 | 3 | 1 | 1 | 1 | 0 | 1 | 1
  Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  None | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Intraoperative Actual Versus Predicted Blood Loss as Assessed by the Operating Surgeon
Description: The predicted blood loss will be estimated preoperatively by the operating surgeon based on a hemostatically normal individual of the same sex, age, stature and co-morbidities as the participant. The actual blood loss will be assessed consisting of the estimated blood loss, including into swabs, towels and suction during the procedure, per the anesthesiologist's record.
Time Frame: Day 0 (at completion of surgery)
Population: For predicted blood loss the number of participants analyzed is 14 as for one participant (included in the major surgery reporting group) the predicted blood loss was not collected. The full analysis data set, including all participants who received investigational product and have at least 1 hemostatic assessment, was used for analysis.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Recombinant Von Willebrand Factor (rVWF) | Minor Surgery | Major Surgery | Oral Surgery | Von Willebrand Disease Type 1 | Von Willebrand Disease Type 2A | Von Willebrand Disease Type 2B | Von Willebrand Disease Type 2M | Von Willebrand Disease Type 3
Number analyzed (Participants) | 15 | 4 | 10 | 1 | 3 | 2 | 1 | 1 | 8
mL
  Actual blood loss | 94.3 (177.88) | 0.0 (0.00) | 127.0 (209.27) | 145.0 (NA) — No standard deviation possible as only one participant was analyzed. | 115.0 (103.32) | 42.5 (53.03) | 50.0 (NA) — No standard deviation possible as only one participant was analyzed. | 50.0 (NA) — No standard deviation possible as only one participant was analyzed. | 110.6 (240.87)
  Predicted blood loss: number analyzed (Participants) | 14 | 4 | 9 | 1 | 3 | 1 | 1 | 1 | 8
  Predicted blood loss | 106.1 (161.82) | 2.5 (5.00) | 152.8 (186.33) | 100.0 (NA) — No standard deviation possible as only one participant was analyzed. | 100.0 (100.00) | 10.0 (NA) — No standard deviation possible as only one participant was analyzed. | 50.0 (NA) — No standard deviation possible as only one participant was analyzed. | 50.0 (NA) — No standard deviation possible as only one participant was analyzed. | 134.4 (206.46)

3. Secondary Outcome: Intraoperative Actual Blood Loss Relative to Predicted Blood Loss
Description: Actual blood loss relative to predicted blood loss will be calculated as [Actual Blood loss (mL)] divided by [Predicted Blood Loss (mL) multiplied by 100.
Time Frame: Day 0 (at completion of surgery)
Population: Number of participants analyzed is 11, as for 3 participants the actual and the predicted blood loss was zero and for 1 participant the predicted blood loss was not collected. Therefore 'actual blood loss relative to predicted blood loss' could not be calculated. The full analysis data set was used for the analysis of this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Recombinant Von Willebrand Factor (rVWF) | Minor Surgery | Major Surgery | Oral Surgery | Von Willebrand Disease Type 1 | Von Willebrand Disease Type 2A | Von Willebrand Disease Type 2B | Von Willebrand Disease Type 2M | Von Willebrand Disease Type 3
Number analyzed (Participants) | 11 | 1 | 9 | 1 | 2 | 1 | 1 | 1 | 6
Percent | 69.6 (44.77) | 0.0 (NA) — No standard deviation possible as only one participant was analyzed. | 68.9 (34.48) | 145.0 (NA) — No standard deviation possible as only one participant was analyzed. | 122.5 (31.82) | 50.0 (NA) — No standard deviation possible as only one participant was analyzed. | 100.0 (NA) — No standard deviation possible as only one participant was analyzed. | 100.0 (NA) — No standard deviation possible as only one participant was analyzed. | 45.0 (38.92)

4. Secondary Outcome: Intraoperative Actual Versus Predicted Blood Loss Score as Assessed by the Operating Surgeon
Description: Hemostatic efficacy will be rated on a scale of excellent - good - moderate - none. Excellent: Intraoperative blood loss was less than or equal to the maximum blood loss expected for the type of procedure performed in a hemostatically normal subject (≤ 100%). Good: Intraoperative blood loss was up to 50% more than the maximum expected blood loss for the type of procedure performed in a hemostatically normal subject (101-150%) Moderate: Intraoperative blood loss was more than 50% of the maximum expected blood loss for the type of procedure performed in a hemostatically normal subject (>150%). None: Uncontrolled hemorrhage that was the result of inadequate therapeutic response despite proper dosing, necessitating a change of clotting factor replacement regimen.
Time Frame: Day 0 (at completion of surgery)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Von Willebrand Factor (rVWF) | Minor Surgery | Major Surgery | Oral Surgery | Von Willebrand Disease Type 1 | Von Willebrand Disease Type 2A | Von Willebrand Disease Type 2B | Von Willebrand Disease Type 2M | Von Willebrand Disease Type 3
Number analyzed (Participants) | 15 | 4 | 10 | 1 | 3 | 2 | 1 | 1 | 8
Participants
  Excellent | 13 | 4 | 8 | 1 | 3 | 1 | 1 | 1 | 7
  Good | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1
  Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  None | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Intraoperative Hemostatic Efficacy Score as Assessed by the Operating Surgeon
Description: Hemostatic efficacy will be rated on a scale of excellent - good - moderate - none. Excellent: Intraoperative hemostasis achieved with rVWF with our without ADVATE was as good or better than that expected for the type of surgical procedure performed in a hemostatically normal subject. Good: Intraoperative hemostasis achieved with rVWF with or without ADVATE was probably as good as that expected for the type of surgical procedure performed in a hemostatically normal subject. Moderate: Intraoperative hemostasis with rVWF with or without ADVATE was clearly less than optimal for the type of procedure performed but was maintained without the need to change the rVWF concentrate. None: Participant experienced uncontrolled bleeding that was the result of inadequate therapeutic response despite proper dosing, necessitating a change of rVWF concentrate.
Time Frame: Day 0 (at completion of surgery)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Von Willebrand Factor (rVWF) | Minor Surgery | Major Surgery | Oral Surgery | Von Willebrand Disease Type 1 | Von Willebrand Disease Type 2A | Von Willebrand Disease Type 2B | Von Willebrand Disease Type 2M | Von Willebrand Disease Type 3
Number analyzed (Participants) | 15 | 4 | 10 | 1 | 3 | 2 | 1 | 1 | 8
Participants
  Excellent | 13 | 4 | 8 | 1 | 3 | 1 | 1 | 1 | 7
  Good | 2 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1
  Moderate | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  None | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Daily Intra- and Postoperative Weight-adjusted Dose of rVWF With or Without ADVATE
Time Frame: Daily, from day of surgery through postoperative Day 14 (± 2 days)
Population: Number of participants analyzed is different for the time points according to individual treatment. The full analysis data set, including all participants who received investigational product and have at least 1 hemostatic assessment, was used for analysis.
Measure: Median (Inter-Quartile Range); unit: IU/kg
Arm/Group | Recombinant Von Willebrand Factor (rVWF)
Number analyzed (Participants) | 15
IU/kg
  intraoperative: number analyzed (Participants) | 1
  intraoperative | 18.1 [18.1 to 18.1]
  postoperative day 1: number analyzed (Participants) | 3
  postoperative day 1 | 23.5 [16.9 to 47.2]
  postoperative day 2: number analyzed (Participants) | 11
  postoperative day 2 | 42.3 [23.2 to 50.6]
  postoperative day 3: number analyzed (Participants) | 12
  postoperative day 3 | 28.6 [20.6 to 48.9]
  postoperative day 4: number analyzed (Participants) | 9
  postoperative day 4 | 33.9 [23.2 to 44.3]
  postoperative day 5: number analyzed (Participants) | 7
  postoperative day 5 | 31.5 [18.8 to 47.2]
  postoperative day 6: number analyzed (Participants) | 5
  postoperative day 6 | 23.2 [18.8 to 23.6]
  postoperative day 7: number analyzed (Participants) | 5
  postoperative day 7 | 23.8 [23.6 to 50.8]
  postoperative day 8: number analyzed (Participants) | 7
  postoperative day 8 | 33.9 [23.6 to 53.6]
  postoperative day 9: number analyzed (Participants) | 3
  postoperative day 9 | 23.6 [16.3 to 53.6]
  postoperative day 10: number analyzed (Participants) | 3
  postoperative day 10 | 23.6 [16.3 to 34.8]
  postoperative day 11: number analyzed (Participants) | 3
  postoperative day 11 | 23.6 [16.3 to 53.6]
  postoperative day 12: number analyzed (Participants) | 4
  postoperative day 12 | 29.3 [20.1 to 44.2]
  postoperative day 13: number analyzed (Participants) | 1
  postoperative day 13 | 16.3 [16.3 to 16.3]
  postoperative day 14: number analyzed (Participants) | 2
  postoperative day 14 | 25.5 [16.3 to 34.8]
  postoperative day 15: number analyzed (Participants) | 1
  postoperative day 15 | 16.3 [16.3 to 16.3]

7. Secondary Outcome: Occurrence of Adverse Events
Description: Treatment emergent adverse events (TEAEs) and treatment emergent serious adverse events (TESAEs) will be evaluated.
Time Frame: From first infusion of investigational product through study completion (ie, 14 (± 2) days post surgery)
Population: The safety analysis data set, including all participants who received any amount of investigational product, was used for analysis of this outcome measure.
Measure: Number; unit: Adverse Events
Arm/Group | Recombinant Von Willebrand Factor (rVWF)
Number analyzed (Participants) | 15
Adverse Events
  Treatment emergent Adverse Events (TEAEs) | 12
  Severe TEAEs | 1
  TEAEs related to rVWF | 0
  TEAEs related to ADVATE | 0
  TEAEs related to both rVWF and ADVATE | 0
  Treatment emergent Serious Adverse Events (TESAEs) | 2
  TESAEs related to rVWF | 0
  TESAEs related to ADVATE | 0
  TESAEs related to both rVWF and ADVATE | 0
  TEAEs leading to discontinuation of rVWF | 0
  TEAEs leading to discontinuation of ADVATE | 0
  TEAEs leading to discontinuation of study | 0
  TEAEs leading to death | 0
  TEAEs related to study procedure | 0
  TESAEs related to study procedure | 0

8. Secondary Outcome: Occurrence of Thrombotic Events
Description: Treatment emergent adverse events (TEAEs) and treatment emergent serious adverse events (TESAEs) will be evaluated for thrombotic events.
Time Frame: From first infusion of investigational product through study completion (ie, 14 (± 2) days post surgery)
Population: as for outcome 7
Measure: Number; unit: Adverse Events
Arm/Group | Recombinant Von Willebrand Factor (rVWF)
Number analyzed (Participants) | 15
Adverse Events
  Thrombotic TEAEs | 2
  Thrombotic TESAEs | 1

9. Secondary Outcome: Occurrence of Severe Allergic Reactions (eg, Anaphylaxis)
Description: Treatment emergent adverse events (TEAEs) and treatment emergent serious adverse events (TESAEs) will be evaluated for severe allergic reactions.
Time Frame: From first infusion of investigational product through study completion (ie, 14 (± 2) days post surgery)
Population: as for outcome 7
Measure: Number; unit: Adverse Events
Arm/Group | Recombinant Von Willebrand Factor (rVWF)
Number analyzed (Participants) | 15
Adverse Events
  Severe allergic reaction TEAEs | 0
  Severe allergic reaction TESAEs | 0

10. Secondary Outcome: Number of Participants Who Developed Inhibitory and Total Binding Antibodies to Von Willebrand Factor (VWF) and Inhibitory Antibodies to Factor VIII (FVIII)
Description: Participants were treated with recombinant van Willebrand Factor (rVWF) with or without ADVATE.
Time Frame: Testing occurred throughout the study at screening, prior PK infusion, pre-surgery, post surgery in case of excessive bleeding or unexplained bleeding, at postoperative day 7 and at study completion visit (ie. 14 (± 2) days post surgery).
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Von Willebrand Factor (rVWF)
Number analyzed (Participants) | 15
Participants
  Development of inhibitory antibodies to VWF | 0
  Development of total binding antibodies to VWF | 1
  Development of inhibitory antibodies to FVIII | 0

11. Secondary Outcome: Number of Participants Who Developed Antibodies to Chinese Hamster Ovary (CHO) Proteins, Mouse Immunoglobulin G (IgG) or Recombinant Furin (rFurin)
Description: Participants were treated with recombinant van Willebrand Factor (rVWF) with or without ADVATE.
Time Frame: as for outcome 10
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Recombinant Von Willebrand Factor (rVWF)
Number analyzed (Participants) | 15
Participants | 0

12. Secondary Outcome: Pharmacokinetics: Area Under the Plasma Concentration Versus Time Curve From 0 to 72 Hours Post-infusion (AUC 0-72 h/Dose)
Description: This assessment is only required for subjects undergoing major surgery. Subjects will receive a PK infusion at a dose of 50±5 IU/kg rVWF:RCo within 42 days prior to surgery. The area under the plasma concentration/time curve from 0 to 72 hours post-infusion will be computed using the linear trapezoidal rule. For the calculation of AUC(0-72h) the levels at 72 hours will be linearly interpolated/extrapolated from the 2 nearest sampling time points. PK analysis was performed for the following analytes: VWF Ristocetin Cofactor Activity (VWF:RCo), VWF Antigen Activity (VWF:Ag), VWF Collagen Binding Activity (VWF:CB), VWF Activity Measured INNOVANCE VWF Ac Assay (VWF:Ac), FVIII Coagulation Activity (FVIII:C)
Time Frame: PK measurements were done within 30 minutes pre-infusion, and post infusion at 30 (± 5) minutes, 60 (± 5) minutes, 6 (± 1) hours, 12 (± 1) hours, 24 (± 2) hours, 48 (± 2) hours and 72 (± 2) hours.
Population: The PK analysis data set, including all participants who underwent PK assessment with data collected at the relevant time points, was used for analysis of this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*IU/dL
Arm/Group | Recombinant Von Willebrand Factor (rVWF)
Number analyzed (Participants) | 11
hours*IU/dL
  VWF:RCo | 31.91 (37.5)
  VWF:Ag | 57.08 (25.6)
  VWF:CB | 63.91 (29.4)
  VWF:Ac | 54.61 (28.1)
  FVIII:C: number analyzed (Participants) | 5
  FVIII:C | 67.49 (31.1)

13. Secondary Outcome: Pharmacokinetics: Area Under the Plasma Concentration Versus Time Curve From Time 0 to Infinity (AUC 0-∞ /Dose)
Description: This assessment is only required for subjects undergoing major surgery. Subjects will receive a PK infusion at a dose of 50±5 IU/kg rVWF:RCo within 42 days prior to surgery. The area under the plasma concentration/time curve from time 0 to infinity and the area under the first moment curve from time 0 to infinity will be calculated as the sum of AUC or AUMC from time 0 to the time of last quantifiable concentration plus a tail area correction calculated as Ct/λz and Ct/λz(t+1/λz), respectively, where Ct is the last quantifiable concentration, t is the time of last quantifiable concentration and λz is the terminal or disposition rate constant. PK analysis was performed for the following analytes: VWF Ristocetin Cofactor Activity (VWF:RCo), VWF Antigen Activity (VWF:Ag), VWF Collagen Binding Activity (VWF:CB), VWF Activity Measured INNOVANCE VWF Ac Assay (VWF:Ac), FVIII Coagulation Activity (FVIII:C)
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*IU/dL
Arm/Group | Recombinant Von Willebrand Factor (rVWF)
Number analyzed (Participants) | 11
hours*IU/dL
  VWF:RCo | 34.43 (43.3)
  VWF:Ag | 68.87 (31.5)
  VWF:CB | 71.82 (34.1)
  VWF:Ac | 61.90 (32.2)
  FVIII:C: number analyzed (Participants) | 3
  FVIII:C | 75.00 (30.9)

14. Secondary Outcome: Pharmacokinetics: Mean Residence Time (MRT)
Description: This assessment is only required for subjects undergoing major surgery. Subjects will receive a PK infusion at a dose of 50±5 IU/kg rVWF:RCo within 42 days prior to surgery. Mean residence time will be calculated as area under the first moment curve from time 0 to infinity divided by the area under the curve time 0 to infinity minus T/2 where T is the duration of the infusion. PK analysis was performed for the following analytes: VWF Ristocetin Cofactor Activity (VWF:RCo), VWF Antigen Activity (VWF:Ag), VWF Collagen Binding Activity (VWF:CB), VWF Activity Measured INNOVANCE VWF Ac Assay (VWF:Ac)
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Recombinant Von Willebrand Factor (rVWF)
Number analyzed (Participants) | 11
hours
  VWF:RCo | 22.69 (41.3)
  VWF:Ag | 37.92 (28.4)
  VWF:CB | 29.35 (31.1)
  VWF:Ac | 29.75 (28.6)

15. Secondary Outcome: Pharmacokinetics: Clearance (CL)
Description: This assessment is only required for subjects undergoing major surgery. Subjects will receive a PK infusion at a dose of 50±5 IU/kg rVWF:RCo within 42 days prior to surgery. Clearance will be calculated as dose (IU/kg) divided by the area under the curve time 0 to infinity. PK analysis was performed for the following analytes: VWF Ristocetin Cofactor Activity (VWF:RCo), VWF Antigen Activity (VWF:Ag), VWF Collagen Binding Activity (VWF:CB), VWF Activity Measured INNOVANCE VWF Ac Assay (VWF:Ac)
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: dL/hour/kg
Arm/Group | Recombinant Von Willebrand Factor (rVWF)
Number analyzed (Participants) | 11
dL/hour/kg
  VWF:RCo | 0.02904 (43.3)
  VWF:Ag | 0.01452 (31.5)
  VWF:CB | 0.01392 (34.1)
  VWF:Ac | 0.01616 (32.2)

16. Secondary Outcome: Pharmacokinetics: Incremental Recovery (IR)
Description: This assessment is only required for subjects undergoing major surgery. Subjects will receive a PK infusion at a dose of 50±5 IU/kg rVWF:RCo within 42 days prior to surgery. Incremental recovery will be calculated as (Cmax minus Cpreinfusion) divided by the dose (IU/kg) where kg refers to the body weight at the time of dosing and Cmax is the observed maximum concentration before correction for pre-infusion values. PK analysis was performed for the following analytes: VWF Ristocetin Cofactor Activity (VWF:RCo), VWF Antigen Activity (VWF:Ag), VWF Collagen Binding Activity (VWF:CB), VWF Activity Measured INNOVANCE VWF Ac Assay (VWF:Ac)
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: IU/dL
Arm/Group | Recombinant Von Willebrand Factor (rVWF)
Number analyzed (Participants) | 11
IU/dL
  VWF:RCo | 1.961 (0.45445)
  VWF:Ag | 1.991 (0.38395)
  VWF:CB | 2.780 (0.56640)
  VWF:Ac | 2.635 (0.38050)

17. Secondary Outcome: Pharmacokinetics: Elimination Phase Half-life (T1/2)
Description: This assessment is only required for subjects undergoing major surgery. Subjects will receive a PK infusion at a dose of 50±5 IU/kg rVWF:RCo within 42 days prior to surgery. Terminal or disposition half-life (T1/2) will be calculated as ln2/λz where λz is the terminal elimination rate constant as calculated in WinNonlin NCA using at least three quantifiable concentrations. PK analysis was performed for the following analytes: VWF Ristocetin Cofactor Activity (VWF:RCo), VWF Antigen Activity (VWF:Ag), VWF Collagen Binding Activity (VWF:CB), VWF Activity Measured INNOVANCE VWF Ac Assay (VWF:Ac)
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Recombinant Von Willebrand Factor (rVWF)
Number analyzed (Participants) | 11
hours
  VWF:RCo | 16.52 (42.7)
  VWF:Ag | 26.88 (26.5)
  VWF:CB | 21.07 (33.2)
  VWF:Ac | 22.19 (28.5)

18. Secondary Outcome: Pharmacokinetics: Volume of Distribution at Steady State (Vss)
Description: This assessment is only required for subjects undergoing major surgery. Subjects will receive a PK infusion at a dose of 50±5 IU/kg rVWF:RCo within 42 days prior to surgery. Vss will be calculated as the clearance multiplied with the mean residence time. PK analysis was performed for the following analytes: VWF Ristocetin Cofactor Activity (VWF:RCo), VWF Antigen Activity (VWF:Ag), VWF Collagen Binding Activity (VWF:CB), VWF Activity Measured INNOVANCE VWF Ac Assay (VWF:Ac)
Time Frame: as for outcome 12
Population: as for outcome 12
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: dL/kg
Arm/Group | Recombinant Von Willebrand Factor (rVWF)
Number analyzed (Participants) | 11
dL/kg
  VWF:RCo | 0.6591 (28.8)
  VWF:Ag | 0.5506 (18.4)
  VWF:CB | 0.4086 (24.0)
  VWF:Ac | 0.4806 (21.5)

ADVERSE EVENTS:
Time Frame: Throughout the study period (from the first exposure to investigational product until study completion or discontinuation date). Total study duration: 1 year and 3 months. Per participant: up to 58 days.
Arm/Group | Recombinant Von Willebrand Factor (rVWF)
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 2/15
Other Adverse Events (participants affected / at risk) | 6/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Von Willebrand Factor (rVWF) (N=15)
Diverticulitis (Infections and infestations) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Recombinant Von Willebrand Factor (rVWF) (N=15)
Acne (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Peripheral swelling (General disorders) | 1 (1)
Nasopharyngitis (Infections and infestations) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreements with PIs may vary per requirements of individual PI, but contain common elements. For this study, PIs are restricted from independently publishing results until completion of the multicenter publication or one year after the conclusion of the study at all sites. Baxalta requires a review of results communication (e.g. for confidential information) >= 30 days prior to submission. Baxalta may request an additional delay of <= 6 months (e.g. for intellectual property protection).